CLINICAL TRIAL: NCT04080063
Title: Biological Markers of Functional Effects of Physical Activity : Aging, Immunometabolism and Frailty Project (VIF-APAS)
Brief Title: Biological Markers of Functional Effects of Physical Activity in an Elderly Population
Acronym: BIO-APAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 19-PP-06
Record Dates: First submitted 2019-08-26; First posted 2019-09-06 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Fragility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- adapted physical activity (Experimental): a personalized care will be offered in terms of adapted physical activity
  Interventions: Other: adapted physical activity

INTERVENTIONS:
Other: adapted physical activity — The study begins with an evaluation of physical strenght and cognitive and psychometric assessment.Then, a personalized care will be offered in terms of adapted physical activity. The evaluation protocol will be performed again to measure the impact of physical activity three months after the first assessment.

SUMMARY:
Circulating biomarkers are promising tools for the early diagnosis of aging-associated pathologies. Inflammation and immunity are associated with the risk of sarcopenia and frailty in elderly patients. The investigators investigate the effect of an adapted physical activity program on the metabolism and function of circulating immune cells and miRNA in frail and non-frail elderly subjects. Induced immune changes are analyzed together with that of motor abilities and of frailty status.

DETAILED DESCRIPTION:
Circulating biomarkers are promising tools for early diagnosis of pathologies associated with aging. Inflammation and immunity are associated with the risk of sarcopenia and frailty in elderly patients. The investigators investigate the effect of an adapted physical activity program on the metabolism and function of circulating immune cells and miRNA in frail and non-frail elderly subjects. The main objective is to establish the link between biological markers of aging (immune cells phenotypes and function, miRNA) and motor capacities alteration/improvement. The secondary objectives are: (1) to characterize the functional and immunometabolic dimensions of frailty from objective indicators; (2) to propose a management system through adapted and individualized physical activity, based on objective indicators; (3) to evaluate the clinical impact of both frailty and its preventative management through physical activity; and (4) to identified new biomarkers of frailty. A total of 100 patients categorized as frail, pre-frail, and non-frail after a standardized geriatric evaluation are included in a comparative and interventional study. Exercise intervention consists in a 12-weeks physical activity program. Blood sample and physical/psychological functional measurements are performed before and after the 12-weeks physical activity program. ANOVA tests and correlational analysis will be performed. The finality of the study is to improve the medical prescription of physical activities in elderly patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient who signed the informed consent
* Older men and women ≥ 65 years
* Can walk without technical help

Exclusion Criteria:

* Patient with protective measures (guardianship, curatorship, and deprivation of liberty).
* Patient with a neurological problem
* No affiliation to a social security scheme (beneficiary or assignee)
* Knee and / or hip prosthesis
* Orthopedic complications with repercussions on walking activities

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 92 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2022-02-21 (Actual); Study Completion 2022-02-21 (Actual)

PRIMARY OUTCOMES:
analysis of phenotype of circulating T cells | change from baseline physical activity at 3 months
  Measurement of T cell populations determined by flow cytometry (FACS) Different antibodies will be used to caracterize different sub-population (CD3+ ; CD4+ ; CD8+ ; T-regulator ; T-helper 1 and 17)
Concentration of mRNAs related to PPARβ/δ gene expression | change from baseline physical activity at 3 months
  Analysis of mRNAs from blood sample related to PPARβ/δ gene expression by Luminex technology

CONTACTS AND LOCATIONS:
Overall Officials: Olivier GUERIN, Principal Investigator — guerin.o@chu-nice.fr
Locations (1):
- CHU de Nice, Nice, France